CLINICAL TRIAL: NCT02536677
Title: The Evaluation and Management of Patients With Acute ChesT Pain in China
Acronym: EMPACT
Status: Completed | Type: Observational
Sponsor: Yuguo Chen (Other)
Collaborators: People's Hospital of Jinxiang County (Unknown); People's Hospital of Chengwu (Unknown); Traditional Chinese Medicine Hospital of Wucheng County (Unknown); People's Hospital of Longkou City (Unknown); People's Hospital of Gaomi City (Unknown); Linyi People's Hospital (Other); People's Hospital of Wenshang County (Unknown); The 2nd People's Hospital of Liaocheng City (Unknown); People's Hospital of Shouguang City (Unknown); Traditional Chinese Medicine Hospital of Pingyin County (Unknown); Traditional Chinese Medicine Hospital of Laoling City (Unknown); The 2nd People's Hospital of Dongying City (Unknown); Affiliated Hospital of Shandong Academy of Medical Sciences (Unknown); People's Hospital of Shizhong District, Jinan City (Unknown); The 2nd People's Hospital of Dezhou City (Unknown); Central Hospital of Zibo (Other); Jining Medical University (Other); People's Hospital of Mudan, Heze City (Unknown); The 3rd People's Hospital of Jinan City (Unknown); Qianfoshan Hospital (Other); Xinlongzhuang Colliery Hospital (Unknown); The 2nd Traditional Chinese Medicine Hospital of Taian City (Unknown); Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor-Investigator, Yuguo Chen, President, Chinese Society of Emergency Medicine;Director, Chest Pain Center, Qilu Hospital of Shandong University, Qilu Hospital of Shandong University
Organization: Qilu Hospital of Shandong University (Other)
Other Study IDs: QLEmer201507
Record Dates: First submitted 2015-08-27; First posted 2015-09-01 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Acute Chest Pain; Acute Coronary Syndrome
Keywords: Acute Chest Pain; Acute Coronary Syndrome; Evaluation and Management; Decision Aid; Healthcare Utilization
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No

SUMMARY:
EMPACT is the first attempt to comprehensively evaluate the current emergency care of acute chest pain from a regional representative sample in China.Findings will allow new opportunities to facilitate the clinical quality improvements and ultimately reduce the mortality and health care burden in patients with acute chest pain. It also will help to establish a regional network and database for further research and performance improvement.

ELIGIBILITY:
Inclusion criteria

1. Eighteen years and older
2. Presenting to the ED
3. With acute chest pain or suspected ACS
4. Symptoms occurring within 24 hours
5. Informed consent from patient or next of kin

Exclusion criteria

1. Chest pain caused by trauma
2. Persisting or recurrent chest pain caused by rheumatic diseases or cancer
3. Transferred from another grade II or grade III hospital
4. Presenting to the ED again within 30 days after initial enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We used a stratified random sampling design to generate a Shandong province representative sample of hospitals. Twenty two hospitals were randomly selected including 12 rural hospitals, 6 grade II and 4 grade III urban hospitals. One grade II-urban hospital refused to participate. As a coordinating center, Qilu Hospital of Shandong University participated in the study without being sampled. Finally, 22 hospitals were included.
  A total of more than 10000 patients were anticipated to be consecutively enrolled from the participating hospitals over the course of the 12-month program. The beginning dates of enrollment in 22 centers were distributed from January, 2016 to September 2016.
Sampling Method: Probability Sample
Enrollment: 8374 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac events (MACE) | 30 days after presenting to the emergency departments(ED)
  The primary outcome was a composite of adjudicated MACEs, including death from all causes, non-fatal acute myocardial infarction (AMI), urgent revascularization, stroke, cardiac arrest, and cardiogenic shock.

SECONDARY OUTCOMES:
revisiting to ED and rehospitalization | 30 days after presenting to the EDs

CONTACTS AND LOCATIONS:
Overall Officials: Yuguo Chen, M.D., Ph.D, Study Chair — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

REFERENCES:
- [Derived] Cheng K, Zheng W, Wang J, Wu S, Zheng J, Sang W, Ma J, Pang J, Pan C, Wang G, Wu Y, Chen Y, Xu F. Incidence, management and outcomes of patients with acute chest pain presenting to the emergency departments in China: findings from a prospective multicentre registry. BMJ Open. 2025 Mar 27;15(3):e091085. doi: 10.1136/bmjopen-2024-091085. PMID 40147987
- [Derived] Yin X, Pan X, Zhang J, Wu S, Cui W, Wang Y, Li C, Wang J, Chen Y. Impact of admission glucose and 30-day major adverse cardiovascular events on patients with chest pain in an emergency setting: insights from the China EMPACT registry. Front Cardiovasc Med. 2024 Oct 9;11:1367704. doi: 10.3389/fcvm.2024.1367704. eCollection 2024. PMID 39444552
- [Derived] Zheng W, Wang J, Xu F, Zheng J, Zhang H, Ma J, Wang G, Wang H, Chew DP, Chen Y. Evaluation and management of patients with acute chest pain in China (EMPACT): protocol for a prospective, multicentre registry study. BMJ Open. 2018 Jan 23;8(1):e017872. doi: 10.1136/bmjopen-2017-017872. PMID 29362251